CLINICAL TRIAL: NCT03897907
Title: The Effect of Psychologically Informed Education in Adolescents With Patellofemoral Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Mitchell Selhorst, Physical Therapist/Principle Investigator, Nationwide Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB18-00724
Record Dates: First submitted 2019-03-29; First posted 2019-04-01 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Patellofemoral Pain Syndrome; Anterior Knee Pain Syndrome
MeSH Terms: conditions — Patellofemoral Pain Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: This research study is a double-blinded randomized controlled trial. The participants will not be made aware which education video they watch is the control and which is the intervention. The study staff will be blinded to group allocation until after measurements are completed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Psychologically Informed Education (Experimental): This arm will provide an education intervention which will attempt to address maladaptive psychological behaviors in adolescents with knee pain
  Interventions: Other: Psychologically Informed Education Video
- Control Education (Placebo Comparator): This arm will provide education of basic knee anatomy and will not address maladaptive psychological behaviors.
  Interventions: Other: Anatomy Education Video

INTERVENTIONS:
Other: Psychologically Informed Education Video — The education session will teach participants how the body processes nociception and experiences pain, and pain does not mean tissues are being damaged. Additionally we will use the framework called the "Common Sense Model of Self-Regulation" which advocates for education to address five cognitive dimensions: (1) identity (the effort to evaluate symptoms and label the illness); (2) cause (the subjectively formulated belief of what is causing the symptoms); (3) time-line (the patient's perception of how long the problem will last); (4) consequences (the patient's predictions of how the illness will affect them in different areas of their life); and (5) controllability (the patient's belief regarding their outcome and personal ability to change it)
  Arms: Psychologically Informed Education
Other: Anatomy Education Video — Participants in the control group will watch three videos equal in length to the psychologically-informed videos. The control videos will discuss anatomy of the lower extremity, basic instruction in proper lower extremity biomechanics, and simple lower extremity exercises. The control videos will provide no psychologically-informed education or positive reinforcement about the condition.
  Arms: Control Education

SUMMARY:
This is a randomized prospective study assessing the impact of psychosocial factors on pain and physical performance among adolescents with anterior knee pain. A set of psychosocial surveys assessing activity-related fear, stress, anxiety and depression will be completed by the participant/parents. Participants will then complete clinical tests of physical performance, numeric pain rating scale, and a self-report questionnaire of functional ability. Participants will then be randomized into one of two psychosocial intervention groups (psychologically informed education group and a control group). After participants receive their assigned education intervention, the clinical tests of pain and self-reported functional ability will be readministered. Participants with anterior knee pain will then complete follow-up surveys of their psychosocial beliefs, pain and self-reported functional ability through REDcap at immediately post-intervention, 2 weeks, 6 weeks, and 3 months.

DETAILED DESCRIPTION:
This study will be a prospective randomized controlled trial design. Participants will complete the randomized intervention immediately after completing baseline testing. Post-intervention testing will also be completed immediately after the randomized intervention. A follow-up REDcap survey will be sent by email to assess function and pain at 2 weeks, 6 weeks and 3 months.

Intervention Psychologically Informed Education Group Psychologically Informed Education Medium There are many ways to provide patient education, but the investigators believe that adolescents will respond well to video education on a tablet. Adolescents are extremely comfortable with this technology, and the video will allow for standardized education among all participants.

Development of Psychologically Informed Education for adolescents with AKP Recommended adult pain science education will be modified using published recommendations for the adolescent population and tailored to anterior knee pain.(Robins, Perron, Heathcote, & Simons, 2016) The education session will teach participants how the body processes nociception and experiences pain, and pain does not mean tissues are being damaged. Additionally the psychologically informed education video will use the framework called the "Common Sense Model of Self-Regulation" which advocates for education to address five cognitive dimensions: (1) identity (the effort to evaluate symptoms and label the illness); (2) cause (the subjectively formulated belief of what is causing the symptoms); (3) time-line (the patient's perception of how long the problem will last); (4) consequences (the patient's predictions of how the illness will affect them in different areas of their life); and (5) controllability (the patient's belief regarding their outcome and personal ability to change it).(Leventhal, Phillips, & Burns, 2016) Control Group Participants in the control education group will watch a video on the iPad equal in length to the psychologically informed education video. The control video will discuss basic anatomy of the knee and provide no psychosocial education or positive reinforcement about their condition.

ELIGIBILITY:
Inclusion Criteria:

Having patellofemoral pain as defined as: Pain around or behind the patella, which is aggravated by at least one activity that loads the patellofemoral joint during weight bearing on a flexed knee (e.g., squatting, stair ambulation, jogging/running, hopping/jumping)

Exclusion Criteria:

1. Prior history of patellar dislocation.
2. Suspicion of other diagnosis of the knee by evaluating physical therapist or principal investigator.
3. Other concomitant injury of the leg.
4. Prior history of knee surgery.
5. Red flags present for non-musculoskeletal involvement (bowel/bladder problems, saddle anesthesia, progressive neurological deficits, recent fever or infection, unexplained weight loss, unable to change symptoms with mechanical testing).
6. Numbness and tingling in any lumbar dermatome.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 68 (Actual)
Dates: Start 2019-04-05 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Change in Anterior Knee Pain Scale | Time Frame: Baseline, 2 weeks (12-16 days post-evaluation), 6 weeks (39-46 days post-evaluation), and 3 months
  Assessment of change of the Anterior Knee Pain Scale (AKPS). The AKPS is a self-reported 13 item questionnaire with discrete categories related to various levels of current knee function. Categories within each item are weighted, and responses are summed to provide an overall score of 0-100, with 100 representing no disability. The Anterior Knee Pain Scale is found to be valid and reliable in patients from 12-50 years of age presenting with anterior knee pain with a test-retest reliability of .95 (Watson, 2005). A change of 10 points represent the minimal clinical difference (Crossley, 2004).

SECONDARY OUTCOMES:
Change in Numeric Pain Rating Scale | Time Frame: Baseline, 2 weeks (12-16 days post-evaluation), 6 weeks (39-46 days post-evaluation), and 3 months
  The Numeric Pain rating scale asks the patient their highest pain in the last 24 hours. The Numeric Pain Rating Scale is a 0-10 scale subjectively assessing a patients perceived level of pain. With 0 on the scale = to no pain, and 10 = to the worst pain imaginable. The use of the Numerical Pain Rating Scale for assessing pain has been validated for use in patients with knee pain and has been found to have a minimal detectable change of 1 points.
Change in Fear-Avoidance Beliefs | Time Frame: Baseline, immediately post-intervention, 2 weeks (12-16 days post-evaluation),
  Fear avoidance beliefs as measured by the Fear Avoidance Beliefs Questionnaire-Physical Activity Subscale
Change in Kinesiophobia | Time Frame: Baseline, immediately post-intervention, 2 weeks (12-16 days post-evaluation),
  Change in kinesiophobia beliefs as measure by the Tampa Scale for Kinesiophobia-11 scale
Change in Pain Catastrophizing | Time Frame: Baseline, immediately post-intervention, 2 weeks (12-16 days post-evaluation),
  Change in pain catastrophizing as measured by the pain catastrophizing scale-child version

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell Selhorst, DPT, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital Sports and Ortho Physical Therapy, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, CSR
Access Criteria: As a part of this research, it will be necessary to collect identifying information. Even though the final dataset will be stripped of identifiers prior to release for sharing, the patient sample is composed of minors who are a protected patient population Thus, we will make the data and associated documentation available to users only under a data-sharing agreement that provides for: (1) a commitment to using the data only for research purposes and not to identify any individual participant; (2) a commitment to securing the data using appropriate computer technology; and (3) a commitment to destroying or returning the data after analyses are completed. Aggregate data including sample means, standard deviations, frequencies and significance values will be shared through peer-reviewed publications and conference abstracts. Email requests for data-sharing agreements to Mitchell.Selhorst@Nationwidechildrens.org

REFERENCES:
- [Background] Grotle M, Garratt AM, Krogstad Jenssen H, Stuge B. Reliability and construct validity of self-report questionnaires for patients with pelvic girdle pain. Phys Ther. 2012 Jan;92(1):111-23. doi: 10.2522/ptj.20110076. Epub 2011 Oct 20. PMID 22016375
- [Background] Leventhal H, Phillips LA, Burns E. The Common-Sense Model of Self-Regulation (CSM): a dynamic framework for understanding illness self-management. J Behav Med. 2016 Dec;39(6):935-946. doi: 10.1007/s10865-016-9782-2. Epub 2016 Aug 11. PMID 27515801
- [Background] Robins H, Perron V, Heathcote LC, Simons LE. Pain Neuroscience Education: State of the Art and Application in Pediatrics. Children (Basel). 2016 Dec 21;3(4):43. doi: 10.3390/children3040043. PMID 28009822
- [Background] Vlaeyen JWS, Linton SJ. Fear-avoidance model of chronic musculoskeletal pain: 12 years on. Pain. 2012 Jun;153(6):1144-1147. doi: 10.1016/j.pain.2011.12.009. Epub 2012 Feb 8. No abstract available. PMID 22321917
- [Background] Wang YC, Hart DL, Stratford PW, Mioduski JE. Baseline dependency of minimal clinically important improvement. Phys Ther. 2011 May;91(5):675-88. doi: 10.2522/ptj.20100229. Epub 2011 Mar 3. PMID 21372203
- [Background] Watson CJ, Propps M, Ratner J, Zeigler DL, Horton P, Smith SS. Reliability and responsiveness of the lower extremity functional scale and the anterior knee pain scale in patients with anterior knee pain. J Orthop Sports Phys Ther. 2005 Mar;35(3):136-46. doi: 10.2519/jospt.2005.35.3.136. PMID 15839307
- [Background] Crossley KM, Bennell KL, Cowan SM, Green S. Analysis of outcome measures for persons with patellofemoral pain: which are reliable and valid? Arch Phys Med Rehabil. 2004 May;85(5):815-22. doi: 10.1016/s0003-9993(03)00613-0. PMID 15129407